CLINICAL TRIAL: NCT04289051
Title: Clinical Evaluation of the Efficacy of an Intra Oral Rinse for Patients With Xerostomia
Brief Title: Clinical Evaluation of Oral Rinse for Xerostomia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunstar Americas (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLP-2020-02-01-1
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Results first posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2021-12

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- HYDRAL Oral Rinse (Experimental): Subjects use the oral rinse four times daily adding to a regular oral hygiene routine with a fluoride toothpaste and a soft tooth brush.
  Interventions: Device: HYDRAL Oral Rinse; Device: BIOTENE® Oral Rinse; Device: Placebo Oral Rinse
- BIOTENE® Oral Rinse (Active Comparator): Subjects use the oral rinse four times daily adding to a regular oral hygiene routine with a fluoride toothpaste and a soft tooth brush.
  Interventions: Device: HYDRAL Oral Rinse; Device: BIOTENE® Oral Rinse; Device: Placebo Oral Rinse
- Placebo Oral Rinse (Placebo Comparator): Subjects use the oral rinse four times daily adding to a regular oral hygiene routine with a fluoride toothpaste and a soft tooth brush.
  Interventions: Device: HYDRAL Oral Rinse; Device: BIOTENE® Oral Rinse; Device: Placebo Oral Rinse

INTERVENTIONS:
Device: HYDRAL Oral Rinse — Application 4 times a day for two weeks
Device: BIOTENE® Oral Rinse — Application 4 times a day for two weeks
Device: Placebo Oral Rinse — Application 4 times a day for two weeks

SUMMARY:
Xerostomia causes a difficulty in eating, have irritated oral tissues, and a poor quality of life. The new oral rinse was designed to reduce the symptoms and improve the patient's quality of life. The objectives of the clinical study is to evaluate the effectiveness of the oral rinse comparing to the placebo product and the control product in the market.

This is a randomized double-blind placebo controlled crossover study with 39 patients receiving treatment. Patients will be randomly allocated to three treatment groups. Patients will use the assigned oral rinse four times a day for two weeks. Dry mouth symptoms and other endpoints will be assessed subjectively and objectively at baseline and Day 14. Patients will be assigned to another treatment after one week wash-out period.

ELIGIBILITY:
Inclusion Criteria:

1. Must have read, understood and signed an informed consent prior to being entered into the study.
2. Must be 18 to 80 years of age, male or female.
3. Have at least 20 natural or restored teeth.
4. Have an unstimulated salivary flow rate <0.20 ml/minute which represents a significant reduction of normal salivary function
5. Must have subjective xerostomia symptom: minimum level of 4 on a 10 centimeters Visual Analog Scale (VAS) [How would you score dryness of your mouth?]
6. Agree not to have a dental prophylaxis or any other elective, non-emergency dental procedures (other than those provided during the study) any time during the study.
7. Agree to abstain from the use of any products for xerostomia other than those provided in the study.
8. Agree to comply with the conditions and schedule of the study.

Exclusion Criteria:

1. Physical limitations or restrictions that might preclude normal tooth brushing.
2. Evidence of gross oral pathology, including widespread caries or chronic neglect, extensive restoration, pre-existing gross plaque or soft or hard tissue tumor of the oral cavity.
3. Presence of severe gingivitis with 30 or more sites showing bleeding on probing.
4. Evidence of major oral hard or soft tissue lesions or trauma at the baseline visit as determined by the Investigator/Examiner.
5. Chronic disease with concomitant oral manifestations other than xerostomia
6. Conditions requiring antibiotic treatment prior to dental prophylaxis and invasive procedures, such as heart murmur, history of rheumatic fever, valvular disease or certain prosthetic implants.
7. History of hepatic or renal disease, uncontrolled diabetes, or other serious conditions or transmittable diseases.
8. Subjects who are currently undergoing, or require, extensive dental work, orthodontic treatment or periodontal surgery or orthodontic treatment in the preceding 3 months
9. Currently using bleaching trays
10. History of radiotherapy, head and neck cancer or Sjogren's syndrome.
11. History of significant adverse effects following use of oral hygiene products such as toothpastes and mouthrinses.
12. Subjects who are nursing, pregnant or plan to become pregnant for the duration of the study.
13. Currently breast feeding
14. Eating disorders
15. Recent history of substance abuse
16. Participation in other clinical studies within 14 days of screening
17. Smoking >10 cigarettes/day
18. Chewing tobacco
19. Daily use of symptom alleviating products against xerostomia within 7 days of screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo, The Center for Dental Studies, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- HYDRAL Oral Rinse - Placebo Oral Rinse - Biotene Oral Rinse: Subjects use following oral rinses four times daily adding to a regular oral hygiene routine with a fluoride toothpaste and a soft tooth brush. One-week washout period separates two different interventions of two weeks.
  First intervention: HYDRAL Oral Rinse Second intervention: Placebo Oral Rinse Third intervention: BIOTENE® Oral Rinse
- Placebo Oral Rinse - Biotene Oral Rinse - HYDRAL Oral Rinse: Subjects use following oral rinses four times daily adding to a regular oral hygiene routine with a fluoride toothpaste and a soft tooth brush. One-week washout period separates two different interventions of 2 weeks.
  First intervention: Placebo Oral Rinse Second intervention: BIOTENE® Oral Rinse Third intervention: HYDRAL Oral Rinse
- BIOTENE Oral Rinse - HYDRAL Oral Rinse - Placebo Oral Rinse: Subjects use following oral rinses four times daily adding to a regular oral hygiene routine with a fluoride toothpaste and a soft tooth brush. One-week washout period separates two different interventions of two weeks.
  First intervention: BIOTENE® Oral Rinse Second intervention: HYDRAL Oral Rinse Third intervention: Placebo Oral Rinse
Period: Overall Study
Arm/Group | HYDRAL Oral Rinse - Placebo Oral Rinse - Biotene Oral Rinse | Placebo Oral Rinse - Biotene Oral Rinse - HYDRAL Oral Rinse | BIOTENE Oral Rinse - HYDRAL Oral Rinse - Placebo Oral Rinse
Started | 13 | 13 | 13
First Intervention (2 Weeks) | 13 | 13 | 11
Washout (1 Week) | 13 | 13 | 11
Second Intervention (2 Weeks) | 13 | 13 | 11
Washout (1 Week) | 13 | 13 | 11
Third Intervention (2 Weeks) | 13 | 13 | 11
Completed | 13 | 13 | 11
Not Completed | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Overall Participants: Subject disposition for all arms
Arm/Group | Overall Participants
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 30
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Change in Dry Mouth Symptom by Visual Analog Scale at 14 Days From Baseline
Description: 100 mm visual analog scale for subjective scoring the level of dry mouth (0 mm: not dry at all, 100 mm: very dry). Change in mm was calculated by subtracting the measurement at 14 days from the measurement at baseline. Higher values of the changes from baseline represent a better outcome.
Time Frame: Baseline, 14 days
Measure: Mean (Standard Deviation); unit: mm
Groups:
- HYDRAL Oral Rinse; Placebo Oral Rinse; BIOTENE® Oral Rinse: Subjects use the oral rinse four times daily adding to a regular oral hygiene routine with a fluoride toothpaste and a soft tooth brush for two weeks.
Arm/Group | HYDRAL Oral Rinse | Placebo Oral Rinse | BIOTENE® Oral Rinse
Number analyzed (Participants) | 37 | 37 | 37
mm | 10.1 (2.5) | 11.6 (3.9) | 13.0 (3.2)

2. Primary Outcome: Change in Dry Mouth Symptoms by Xerostomia Questionnaire at 14 Days From Baseline
Description: Questionnaire to assess xerostomia symptoms. Subjects were asked the degree (grade 0: no problems to grade 3: the worst possible problem) of hoarse voice, oral dryness, oral pain, swallowing, and taste loss from which they were suffering in the xerostomia questionnaire. The symptoms scores were summed to calculate a total score per each subject (minimum total score: 0, maximum total score: 15). The change was calculated by subtracting the total score at 14 days from the total score at baseline. Higher values of the changes represent a better outcome (minimum change: -15, maximum change: 15).
Time Frame: Baseline, 14 days
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | HYDRAL Oral Rinse | Placebo Oral Rinse | BIOTENE® Oral Rinse
Number analyzed (Participants) | 37 | 37 | 37
Score on a scale | 1.0 (2.8) | 0.4 (1.7) | 0.5 (1.5)

3. Secondary Outcome: Change in Oral Functions by Revised Oral Assessment Guide at 14 Days From Baseline
Description: Assessment of oral functions by a dental professional. Eight categories were included in the assessment guide: voice, lips, mucous membranes, tongue, gums, teeth, saliva, and swallowing. Each category was described and rated from healthy (score 1) to severe (score 3). Scores for the categories were summed to calculate a total score per each subject (minimum total score: 8, maximum total score: 24). The change was calculated by subtracting the total score at 14 days from the total score at baseline. Higher values of the changes represent a better outcome (minimum change: -16, maximum change: 16).
Time Frame: Baseline, 14 days
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | HYDRAL Oral Rinse | Placebo Oral Rinse | BIOTENE® Oral Rinse
Number analyzed (Participants) | 37 | 37 | 37
Score on a scale | 2.0 (1.3) | 0 (1.7) | 1.2 (1.5)

4. Secondary Outcome: Change in Unstimulated Saliva Flow Rate at 14 Days From Baseline
Description: Unstimulated whole saliva was collected over a 5-minute time period and the volume was measured. Change in mL per minute was calculated by subtracting the measurement at baseline from the measurement at 14 days.
Time Frame: Baseline, 14 days
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | HYDRAL Oral Rinse | Placebo Oral Rinse | BIOTENE® Oral Rinse
Number analyzed (Participants) | 37 | 37 | 37
mL/min | 0.08 (0.11) | 0.00 (0.08) | 0.05 (0.12)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | HYDRAL Oral Rinse | Placebo Oral Rinse | BIOTENE® Oral Rinse
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 2/37 | 2/37 | 6/37
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HYDRAL Oral Rinse (N=37) | Placebo Oral Rinse (N=37) | BIOTENE® Oral Rinse (N=37)
Oral mucosal irritation (Gastrointestinal disorders) | 1 (3) | 2 (4) | 5 (5)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT04289051/Prot_SAP_000.pdf